CLINICAL TRIAL: NCT03941210
Title: Micro RNA as Prediction and/or Prognostic Markers of IRIS in TB-HIV Co-infected Patients
Acronym: miRNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12358
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: HIV Infection; Tuberculosis Infection
Keywords: microRNA; HIV; Tuberculosis; IRIS; Biomarkers
MeSH Terms: conditions — HIV Infections; Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma/cells samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HIV+/TB+: Frozen samples and data from participants recruited in the ANRS 12095 CAMELIA clinical trial and the ANRS 12153 CAPRI NK study will be used for this study arm
  All plasma samples were collected before any treatment during IRIS diagnosis and at W8 post TB treatment initiation
  Interventions: Other: Detection of molecular Biomarkers
- HIV+/TB-: Participants included in this study arm will be HIV+ and TB-
  One time collection of 5 ml of blood will be drawn in EDTA tube for each patient before starting cART and sent to the laboratory for protocol analysis
  Interventions: Other: Detection of molecular Biomarkers
- HIV-/TB+: Participants included in this study arm will be HIV- and TB+
  Collection of 5 ml of blood drawing in EDTA tube will be requested for each patient before starting TB drug treatment and after week 2 and 8 of treatment
  Interventions: Other: Detection of molecular Biomarkers
- HIV-/TB-: Participants included in this study arm will be HIV- and TB-
  Clinical examination to rule out overt evidence of TB and, whenever needed, routine TB testing as per national guidelines (sputum smear ± chest X-ray) in case of symptoms/clinical manifestations suggestive of TB.
  Interventions: Other: Detection of molecular Biomarkers

INTERVENTIONS:
Other: Detection of molecular Biomarkers — MicroRNA expression profile analysis by flow cytometry

SUMMARY:
The role of miRNAs in HIV disease is yet to be completely defined. Host miRNAs target certain HIV genes, thus can affect HIV replication and participate in viral control. miRNAs can also block HIV production through disruption of Gag assembly on cell membranes. miRNA expression can characterize HIV disease phenotype, as has been shown in HIV elite controllers who have a well-defined miRNA expression profile. However, the studies of miRNA in acute infection and co-infections like tuberculosis are lacking. The investigators showed that during immune reconstitution syndrome (IRIS) in HIV/TB coinfected patients, innate immune response play a role as through NK cell degranulation, therefore testing for this could be used as a predictive marker of IRIS.

One of the limitations of miRNA detection is the technique, which is time-consuming, and needs laboratories that are specialized and equipped for molecular biology techniques. In contrast, flow cytometry has been developed in routine labs and has well-standardized techniques. For the routine detection of miRNA, flow cytometry could be the best way to perform high throughput screening for clinical applications.

Flow cytometry is a simple and effective way to evaluate miRNAs expression. In this project the investigators propose to evaluate, using flow cytometry, whether circulating miRNA pattern might be applicable as potential biomarkers in prediction and prognosis of IRIS in HIV/TB co-infected patients. The investigators propose to study the miRNA expression profile in a cohort of patients with a HIV infection and Tuberculosis and correlate it with their clinical evolution. As controls, the investigators propose to analyze expression of miRNAs in healthy controls as well as TB and HIV mono-infected patients.

AIMS OF THE PROPOSAL

1. Identify miRNA expression profile as potential novel predictive and prognostic biomarkers for IRIS.
2. Identify the miRNA expression profile in HIV patients, in TB patients and in HIV/TB co-infected patients.

ELIGIBILITY:
For HIV+/TB+ participants:

Inclusion Criteria

* cf the CAMELIA clinical trial (NCT00226434)

Exclusion Criteria:

* cf the CAMELIA clinical trial (NCT00226434)

For HIV+/TB- participants:

Inclusion Criteria

* Age ≥ 18 years
* HIV+
* CD4 cell count ≤ 200 x 106 cells/l
* No evidence of tuberculosis infection.

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* CD4 cell count > 200 x 106 cells/l
* Evidence of tuberculosis infection
* Non ART naive at inclusion

For HIV-/TB+ participants:

Inclusion Criteria

* Age ≥ 18 years
* HIV-
* Confirmed tuberculosis infection.

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* AFB negative or MTB/RIF negative for MTB,
* History of TB infection
* HIV+

For HIV-/TB- participants:

Inclusion Criteria

* Age ≥ 18 years
* HIV-
* No evidence of tuberculosis infection.

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* Evidence of tuberculosis infection
* HIV+

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 74 TB - HIV co-infected patients (37 TB-IRIS and 37 non TB-IRIS) whose plasma were stored during the ANRS 12095 CAMELIA clinical trial (NCT00226434) and ANRS 12153 CAPRI NK study will be included in the study.
  2. 20 HIV ART naïve patients will be enrolled in Sihanouk Hospital Center of HOPE in Cambodia.
  3. 20 newly active tuberculosis patients will be enrolled in Sihanouk Hospital Center of HOPE in Cambodia.
  4. 20 healthy individuals will be recruited from the patients coming to Pasteur Institute in Cambodia for pre-marital test for HIV and who agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
miRNA expression profile in a cohort of patients with a HIV infection and Tuberculosis and correlate it with their clinical evolution | March 1st 2018 - March 1st 2020
  Evaluate, using flow cytometry, whether circulating miRNA (in plasma and/or exosomes) pattern might be applicable as potential biomarkers in prediction and prognosis of IRIS in HIV/TB co-infected patients.
  Description of miRNA expression profile in a cohort of patients with a HIV infection and Tuberculosis and correlate it with their clinical evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pasteur du Cambodge, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No